CLINICAL TRIAL: NCT06012656
Title: Prospective, Multricentre, Non Controlled, Non-randomized, Open Study for the Evaluation of the Cementless Anatomic Femoral Stem MiniMAX
Brief Title: Prospective Study for the Evaluation of the Cementless Anatomic Femoral Stem Minimax -Launay
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.005.10
Record Dates: First submitted 2023-07-26; First posted 2023-08-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Primary Osteoarthritis; Secondary Osteoarthritis; Traumatic Arthritis; Rheumatoid Arthritis; Congenital Hip Dysplasia; Avascular Necrosis; Fracture; Femur, Head
MeSH Terms: conditions — Arthritis, Rheumatoid; Hip Dislocation, Congenital; Osteonecrosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: MiniMAX — Total or Partial Hip Arthroplasty

SUMMARY:
This is a post-marketing surveillance on MiniMAX Stem

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a clinical condition requiring THA
2. Patient receiving a MiniMAX® stem
3. Patient aged more than 18 years
4. Patient having a Social Insurance or a similar protection regime
5. Patient eligible for an AMIS procedure
6. Patient able to follow the study requirements
7. Patients who are willing to give informed written consent

Exclusion Criteria:

1. Patient with local or systemic infection
2. Participation to biomedical research
3. Patient whose BMI exceeds 40
4. Patient with less than 18 years
5. Protected adults
6. Vulnerable person according to article L1121-6 of the Code de la Santè Publique.
7. Pregnant or lactating woman
8. Patient unable to express his/ her opinion about the participation to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size of 100 patients has been defined based on the literature data to guarantee a sufficient number of patients for the evaluation of the performance of the prosthesis, taking into account a 10% of lost patients (dead or lost at follow-up).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2031-01-02 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | 10 years
  Kaplan Meier method

SECONDARY OUTCOMES:
Functional evaluation | Pre-op, 3 months, 1, 3, 5, 10 years
  Harris Hip Score (HHS): the HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Evaluation of patient satisfaction | Pre-op, 3 months, 1, 3, 5, 10 years
  HOOS (hip disability and osteoarthritis outcome score) questionnaire: HOOS is a questionnaire intended to be used to assess patient's opinion about their hip and associated problems, and to evaluate their symptoms and functional limitations during a therapeutic process.The interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Evaluation of the stem fixation | Pre-op, 3 months, 1, 3, 5, 10 years
  Radiographic evaluation to assess the osteointegration of the stem, the implant positioning, radiolucent lines.
Evaluation of the general and thigh pain | Pre-op, 3 months, 1, 3, 5, 10 years
  Echelle Visuelle Analogique (EVA) and pain location. Interpretation of the EVA scale: no pain 0, low pain 1-3, moderate pain 4-6, severe pain 7-9, extreme pain 10.
Incidence of adverse events | Surgery, Immediate post-op, 3 months, 1, 3, 5, 10 years
  Intraoperative and postoperative complications
Evaluation of the stability of the stem | Pre-op, 3 months, 1, 3, 5, 10 years
  Radiographic evaluation to assess the osteointegration of the stem, the implant positioning, radiolucent lines.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Clinical Angouleme Soyaux, Soyaux, France, France

IPD SHARING:
Plan to Share IPD: No